CLINICAL TRIAL: NCT01371994
Title: A Randomized, Double-Blind, Parallel, Placebo-Controlled, Phase 4, Multicenter Study to Assess Efficacy and Safety of VESIcare® (Solifenacin Succinate) to Improve Urinary Continence of Subjects After Robotic Assisted Radical Prostatectomy
Brief Title: A Study to Assess Efficacy and Safety With Solifenacin Succinate to Improve Urinary Continence After Robotic Assisted Radical Prostatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 905-UC-050
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Urinary Incontinence
Keywords: Radical Robotic Arm; Vesicare; Post Prostatectomy Incontinence; YM905
MeSH Terms: conditions — Urinary Incontinence | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solifenacin succinate (Experimental): Participants received 5 mg solifenacin succinate tablets once a day for 12 weeks. At week 4, based on efficacy and safety and in agreement with the investigator, the dose might be increased to 10 mg (2 tablets of 5 mg) once daily.
  Interventions: Drug: solifenacin succinate
- Placebo (Placebo Comparator): Participants received matching placebo tablets once a day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: solifenacin succinate — oral
  Other Names: Vesicare; YM905
  Arms: Solifenacin succinate
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 12 weeks of treatment of solifenacin succinate versus placebo in participants who are incontinent after Robotic Assisted Radical Prostatectomy.

This study will also assess the effect of 12 weeks of treatment with solifenacin succinate versus placebo on quality of life (QOL) as measured by questionnaires.

DETAILED DESCRIPTION:
The study duration includes a 14-day treatment free wash-out period. The maximum total study duration is 15 weeks (2-3 week screening/washout period and a 12 week treatment period). The Baseline, Week 4, and Week 8 visits will be telephone contact visits.

Participants will complete an electronic daily pad use diary during the study

duration. Participants will also be asked to complete several questionnaires during the study.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Willing and able to complete the daily pad use diary,

American Urology Association Symptom Score (AUASS) with Bother Score, the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF), and the Work Productivity and Activity Impairment Questionnaire (WPAI)

* Has not used any medication for over-active bladder symptoms for at least 14 days prior to enrollment
* Diagnosed with prostate cancer, treated by Robotic Assisted Radical Prostatectomy, is voiding spontaneously and has urinary incontinence one week after removal of the indwelling catheter which requires management with 2 to 10 pads inclusive per day (24 hour days) for 7 consecutive days

Exclusion Criteria:

* Evidence of severe neurologic damage post-prostatectomy
* Evidence of chronic urologic inflammation such as interstitial cystitis and bladder stone; uncontrolled narrow angle glaucoma; urinary or gastric retention or neurogenic bladder
* Symptomatic for urinary tract infection or has a urine culture result which requires treatment as determined by the investigator.
* Clinically significant history of hepatic or renal impairment (2 X Upper Limit of Normal (ULN) values in alanine aminotransferase (ALT), aspartate aminotransferase (AST) or creatinine clearance < 30 ml/min)
* History of diagnosed gastrointestinal obstruction disease
* Any prior history of local radiation therapy to the prostate or rectum or any prior hormonal therapy or has planned such therapy during study conduct
* Known or suspected hypersensitivity to solifenacin succinate, any components, or other anticholinergics
* Treated with any investigational drug within last 30 days
* History of a clinically significant illness or medical condition that would preclude participation in the study
* Diagnosed with New York Heart Association Class III and IV heart failure
* Any of the following peri-operative laboratory results: ALT > 2.0 ULN, AST > 2.0 ULN, serum creatinine > 1.5 mg/L, blood glucose > 130 mg/dL, blood urea nitrogen (BUN) > 23 mg/dL.
* Severe hypertension on peri-operative evaluation which is defined as a sitting systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg, and which is not corrected
* Electrolytes (sodium, potassium, chloride or bicarbonate) that are not in normal range and clinically significant as determined by the investigator in the perioperative period. Can be eligible if electrolytes are corrected to within normal range prior to randomization
* Participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half lives, whichever is longer, prior to the initiation of Screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2011-08-02 (Actual); Primary Completion 2013-10-21 (Actual); Study Completion 2013-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (60):
- United States (58):
  - Urology Centers of Alabama, Homewood, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - University of California, San Diego Moores Cancer Center, La Jolla, California
  - Tower Urology, Los Angeles, California
  - Radiological Associates of Sacramento Medical Group, Inc., Sacramento, California
  - Urology Center of Colorado, Denver, Colorado
  - Urology Associates, Englewood, Colorado
  - Advanced Urology, Parker, Colorado
  - Connecticut Clinical Research Center, Middlebury, Connecticut
  - Grove Hill Medical Center, New Britain, Connecticut
  - Urologic Surgeons of Washington, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Urology Research Network, Hialeah, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Winter Park Urology Associates, Orlando, Florida
  - Southeastern Research Group, Tallahassee, Florida
  - Northwestern University, Chicago, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Northeast Indiana Research, Fort Wayne, Indiana
  - Urology of Indiana, Greenwood, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The Iowa Clinic, West Des Moines, Iowa
  - Tulane University School of Medicine, Department of Urology, New Orleans, Louisiana
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Adult and Pediatric Urology Group, Sartell, Minnesota
  - Five Valley Urology, Missoula, Montana
  - South Nevada Aids Research, Las Vegas, Nevada
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Delaware Valley Urology, Mount Laurel, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Community Care Physicians PC, Albany, New York
  - Brooklyn Urology Research Group, Brooklyn, New York
  - University Urology Associates, New York, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - University of Rochester Medical Center, Rochester, New York
  - AMP Urology, Syracuse, New York
  - Cary Urology, Cary, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Romius Institute of Northwest Ohio, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Pharma Resources, East Providence, Rhode Island
  - Academic Urologists, Chattanooga, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Southeast Urology Network, Memphis, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Methodist Hospital Research Institute, Houston, Texas
  - Methodist Urology Associates, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Urology Group, Seattle, Washington
  - CAMC Institute Clinical Trial Center, Charleston, West Virginia
  - University of Wisconsin Hospital, Madison, Wisconsin
- Canada (2):
  - The Prostate Centre, Diamond Health Care Centre, Vancouver, British Columbia
  - University Health Network/ Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of male patients > 18 years of age who were diagnosed with prostate cancer, treated by robotic assisted radical prostatectomy (RARP) and had urinary incontinence for 1 week following removal of the indwelling catheter.
Pre-assignment Details: Participants meeting the Baseline criteria were randomized 1:1 to 5 mg solifenacin succinate or matching placebo.
Period: Overall Study
Arm/Group | Placebo | Solifenacin Succinate
Started | 320 | 320
Received Treatment | 310 | 313
Completed | 263 | 278
Not Completed | 57 | 42
Not completed — Adverse Event | 3 | 6
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 24 | 17
Not completed — Randomized but Never Received Study Drug | 6 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Miscellaneous Reasons | 6 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set, defined as all participants who took at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Solifenacin Succinate | Total
Number analyzed (Participants) | 310 | 313 | 623
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (6.72) | 60.5 (7.21) | 60.9 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 310 | 313 | 623
Race/Ethnicity, Customized [Number; unit: participants]
  White | 263 | 266 | 529
  Black | 43 | 44 | 87
  Asian | 2 | 3 | 5
  Other | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 284 | 284 | 568
  Hispanic or Latino | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Time From First Dose to Urinary Continence
Description: Urinary continence is defined as the first of three consecutive 24-hour days in which a participant uses no pads, or a pad for security which remains completely dry, during the 12-week treatment period. Participants recorded their daily pad usage in an electronic diary. Kaplan-Meier curves were used to estimate the distribution of cumulative incidence of urinary continence over the 12-week study treatment period. Participants who did not experience the event during the 12-week treatment period were considered as censored at the End of Treatment (EOT) visit or Week 12, whichever occurs first.
Time Frame: 12 weeks
Population: Full analysis set defined as all randomized participants who took at least one dose of study drug and had at least one efficacy endpoint evaluation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 309 | 313
days | NA [93.0 to NA] — Data were not observed during 12-week treatment period due to low incidence of continence events. | NA [NA to NA] — Data were not observed during 12-week treatment period due to low incidence of continence events.
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; The treatment difference in the primary efficacy variable was tested using a log-rank test stratified by (pooled) center and by Baseline daily pad usage (≤3 and >3) at a 2-sided significance level of 0.05; Test type: Superiority or Other; p = 0.1745, Log Rank; Based on a Log-rank test stratified by (pooled) center and Baseline daily pad usage (≤ 3 and > 3)

2. Secondary Outcome: Percentage of Participants Who Gain Continence During 12-week Treatment Period
Description: Urinary continence is defined as three consecutive 24-hour days in which a participant uses no pads or a pad for security which remains completely dry. Participants recorded their daily pad usage in an electronic diary during the 12-week treatment period. End of treatment is the last on-treatment assessment during the treatment period.
Time Frame: Weeks 4, 8, and 12
Population: Full analysis set; the calculation of percentage of participants uses the full analysis set as the denominator at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 309 | 313
percentage of participants
  Week 4 | 10.4 | 11.8
  Week 8 | 18.8 | 21.1
  Week 12 | 19.1 | 26.5
  End of Treatment | 21.4 | 29.1
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 4; Test type: Superiority or Other; p = 0.4833, Cochran-Mantel-Haenszel; Cochran-Mental-Haenszel test stratified by (pooled) center
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 8; Test type: Superiority or Other; p = 0.5761, Cochran-Mantel-Haenszel; Cochran-Mental-Haenszel test stratified by (pooled) center
Statistical Analysis 3: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.0592, Cochran-Mantel-Haenszel; Cochran-Mental-Haenszel test stratified by (pooled) center
Statistical Analysis 4: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.0390, Cochran-Mantel-Haenszel; Cochran-Mental-Haenszel test stratified by (pooled) center

3. Secondary Outcome: Average Daily Pad Usage at Baseline
Description: Participants recorded their daily pad usage in an electronic diary during the 12-week treatment period. A 7-day window was used to calculate the average daily pad usage.
Time Frame: Baseline (7 days prior to Day 1)
Population: Full analysis set with available pad usage data at Baseline.
Measure: Mean (Standard Deviation); unit: pads
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 309 | 313
pads | 5.0 (2.30) | 4.7 (2.16)

4. Secondary Outcome: Change From Baseline in Average Daily Pad Usage
Description: Participants recorded their daily pad usage in an electronic diary during the 12-week treatment period. A 7-day window was used to calculate the average daily pad usage. End of treatment is the last on-treatment assessment during the treatment period.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: Full analysis set with available pad usage data at both Baseline and each time point; "n" indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 298 | 302
pads
  Week 4 (n=297, 302) | -1.9 (0.10) | -2.0 (0.09)
  Week 8 (n=280, 292) | -2.5 (0.10) | -2.8 (0.10)
  Week 12 (n=226, 226) | -3.1 (0.10) | -3.4 (0.10)
  End of treatment (n=298, 302) | -2.9 (0.09) | -3.2 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 4; Test type: Superiority or Other; p = 0.3604, ANCOVA; Based on an analysis of variance model including treatment and (pooled) center as fixed factors; Treatment Difference = 0.1, 95% CI 2-sided [-0.14 to 0.38], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 8; Test type: Superiority or Other; p = 0.0761, ANCOVA; Based on an analysis of variance model including treatment and (pooled) center as fixed factors; Treatment Difference = 0.2, 95% CI 2-sided [-0.03 to 0.52], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.0149, ANCOVA; Based on an analysis of variance model including treatment and (pooled) center as fixed factors; Treatment Difference = 0.4, 95% CI 2-sided [0.07 to 0.64], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.0325, ANCOVA; Based on an analysis of variance model including treatment and (pooled) center as fixed factors; Treatment Difference = 0.3, 95% CI 2-sided [0.02 to 0.52], Standard Error of Mean 0.13

5. Secondary Outcome: American Urology Association Symptom Score (AUASS) at Baseline
Description: Quality of life was measured by the American Urology Association Symptom Score (AUASS). The AUASS includes 7 questions addressing symptoms of frequency, urgency, nocturia (waking during the night to urinate), hesitancy, weak urinary, incomplete emptying, and intermittence. The questionnaire asked participants to consider how these symptoms affected them over the past month on a scale from 0 (not at all) to 5 (almost always). The AUASS is a sum of the 7 symptom scores and ranges from 0 (best) to 35 (worst).
Time Frame: Baseline
Population: Full analysis set with available AUASS data at Baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 306 | 311
units on a scale | 16.7 (7.07) | 16.2 (7.22)

6. Secondary Outcome: Change From Baseline in American Urology Association Symptom Score (AUASS)
Description: Quality of life was measured by the American Urology Association Symptom Score (AUASS). The AUASS includes 7 questions addressing symptoms of frequency, urgency, nocturia (waking during the night to urinate), hesitancy, weak urinary, incomplete emptying, and intermittence. The questionnaire asked participants to consider how these symptoms affected them over the past month on a scale from 0 (not at all) to 5 (almost always). The AUASS Symptom Score is a sum of the 7 symptom scores and ranges from 0 (best) to 35 (worst). End of treatment is the last on-treatment assessment during the treatment period.
Time Frame: Baseline and Week 12
Population: Full analysis set with available AUASS data at both Baseline and each time point; "n" indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 293 | 307
units on a scale
  Week 12 (n=262, 277) | -7.7 (0.33) | -8.0 (0.32)
  End of treatment (n=293, 307) | -7.4 (0.31) | -7.7 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.5186, ANCOVA; Based on an analysis of covariance (ANCOVA) model including Baseline value as a covariates and fixed effects for (pooled) center and treatment; Treatment Difference = 0.3, 95% CI 2-sided [-0.60 to 1.19], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.4521, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 0.3, 95% CI 2-sided [-0.52 to 1.17], Standard Error of Mean 0.43

7. Secondary Outcome: American Urology Association Quality of Life (QOL) Score at Baseline
Description: The American Urology Association (AUA) includes a single bother question which asked participants how they would feel if they had to live with their urinary condition the way it is now for the rest of their life. The bother question score ranges from 0 (delighted) to 6 (terrible).
Time Frame: Baseline
Population: Full analysis set with available AUA QOL data at Baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 306 | 310
units on a scale | 4.8 (1.22) | 4.7 (1.25)

8. Secondary Outcome: Change From Baseline in American Urology Association Quality of Life (QOL) Score
Description: The American Urology Association (AUA) includes a single bother question which asked participants how they would feel if they had to live with their urinary condition the way it is now for the rest of their life. The bother question score ranges from 0 (delighted) to 6 (terrible). End of treatment is the last on-treatment assessment during the treatment period.
Time Frame: Baseline and Week 12
Population: Full analysis set with available AUA data at both Baseline and each time point; "n" indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 292 | 306
units on a scale
  Week 12 (n=261, 276) | -1.9 (0.10) | -2.1 (0.10)
  End of treatment (n=292, 306) | -1.8 (0.09) | -2.0 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.1493, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 0.2, 95% CI 2-sided [-0.07 to 0.47], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.1499, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 0.2, 95% CI 2-sided [-0.07 to 0.44], Standard Error of Mean 0.13

9. Secondary Outcome: International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) QOL Score at Baseline
Description: The ICIQ-SF is a validated self-administered questionnaire designed for patients with urinary incontinence. The ICIQ-SF assessed urinary incontinence using 3 scored questions which ask patients about their frequency of urine leakage, how much urine leakage, and perceived impact of leakage on daily lives over the past 4 weeks. The ICIQ-SF is a sum of the 3 scores and ranges from 0 (low bother) to 21 (maximum bother).
Time Frame: Baseline
Population: Full analysis set with available ICIQ-SF QOL data at Baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 306 | 311
units on a scale | 14.1 (4.10) | 13.8 (4.11)

10. Secondary Outcome: Change From Baseline in International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) QOL Score
Description: as for outcome 9
Time Frame: Baseline and Week 12
Population: Full analysis set with available ICIQ-SF data at both Baseline and each time point; "n" indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 292 | 307
units on a scale
  Week 12 (n=262, 277) | -5.7 (0.26) | -6.2 (0.25)
  End of treatment (n=292, 307) | -5.5 (0.25) | -6.0 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.1279, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 0.5, 95% CI 2-sided [-0.16 to 1.23], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.1038, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 0.6, 95% CI 2-sided [-0.11 to 1.23], Standard Error of Mean 0.34

11. Secondary Outcome: Baseline Work Productivity and Activity Impairment (WPAI): Percent Work Time Missed
Description: Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI asks participants about the effect of urinary leakage on their ability to perform their work-related functions and carry out daily activities over the past seven days. Percent work time missed is derived from the number of hours of work missed due to urinary leakage as a percentage of total hours that should have been worked. A higher percentage indicates more hours missed.
Time Frame: Baseline
Population: Full analysis set participants who were employed prior to the study and with available WPAI data at Baseline.
Measure: Mean (Standard Deviation); unit: percent work time missed
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 96 | 112
percent work time missed | 43.6 (46.22) | 37.9 (45.50)

12. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Work Time Missed
Description: Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI asks participants about the effect of urinary leakage on their ability to perform their work-related functions and carry out daily activities over the past seven days. Percent work time missed is derived from the number of hours of work missed due to urinary leakage as a percentage of total hours that should have been worked. A higher percentage indicates more hours missed. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set including participants who were employed prior to the study and with available WPAI data at both Baseline and each time point; "n" indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: Percent work time missed
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 88 | 102
Percent work time missed
  Week 12 (n= 81, 88) | -37.9 (1.51) | -37.6 (1.42)
  End of treatment (n=88, 102) | -36.8 (2.25) | -34.4 (2.04)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.8876, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = -0.3, 95% CI 2-sided [-4.19 to 3.63], Standard Error of Mean 1.98
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.3950, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = -2.4, 95% CI 2-sided [-8.10 to 3.21], Standard Error of Mean 2.86

13. Secondary Outcome: Baseline Work Productivity and Activity Impairment (WPAI): Percent Impairment While Working
Description: Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI asks participants about the effect of urinary leakage on their ability to perform their work-related functions and carry out daily activities over the past seven days. Percent impairment while working was derived from the participant's assessment of the degree to which urinary leakage affected their productivity while working. A higher percentage indicates greater impairment and less productivity.
Time Frame: Baseline
Population: Full analysis set participants who were employed prior to the study and with available WPAI data at Baseline.
Measure: Mean (Standard Deviation); unit: percent impairment while working
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 75 | 101
percent impairment while working | 35.5 (30.05) | 34.1 (29.70)

14. Secondary Outcome: Change From Baseline in Work Productivity Assessment Index (WPAI): Percent Impairment While Working
Description: Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI asks participants about the effect of urinary leakage on their ability to perform their work-related functions and carry out daily activities over the past seven days. Percent impairment while working was derived from the participant's assessment of the degree to which urinary leakage affected their productivity while working. A higher percentage indicates greater impairment and less productivity. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: percent impairment while working
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 72 | 91
percent impairment while working
  Week 12 (n=66, 80) | -21.8 (1.89) | -23.8 (1.71)
  End of treatment (n=72, 91) | -20.8 (1.96) | -21.8 (1.72)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.4126, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 2.0, 95% CI 2-sided [-2.82 to 6.81], Standard Error of Mean 2.43
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.6959, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 1.0, 95% CI 2-sided [-3.92 to 5.85], Standard Error of Mean 2.47

15. Secondary Outcome: Baseline Work Productivity and Activity Impairment (WPAI): Percent Overall Work Impairment
Description: Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI asks participants about the effect of urinary leakage on their ability to perform their work-related functions and carry out daily activities over the past seven days. Percent overall work impairment takes into account both hours missed due to urinary leakage and the participant's assessment of the degree to which urinary leakage affected their productivity while working. A higher percentage indicates greater impairment and less productivity.
Time Frame: Baseline
Population: Full analysis set participants who were employed prior to the study and with available WPAI data at Baseline.
Measure: Mean (Standard Deviation); unit: percent overall work impairment
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 69 | 89
percent overall work impairment | 42.5 (35.26) | 44.8 (33.41)

16. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Overall Work Impairment
Description: Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI asks participants about the effect of urinary leakage on their ability to perform their work-related functions and carry out daily activities over the past seven days. Percent overall work impairment takes into account both hours missed due to urinary leakage and the participant's assessment of the degree to which urinary leakage affected their productivity while working. A higher percentage indicates greater impairment and less productivity. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: percent overall work impairment
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 65 | 79
percent overall work impairment
  Week 12 (n= 59, 69) | -30.4 (2.18) | -33.7 (1.94)
  End of treatment (n=65, 79) | -30.0 (2.23) | -31.1 (1.95)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.2402, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 3.3, 95% CI 2-sided [-2.26 to 8.91], Standard Error of Mean 2.81
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.6980, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 1.1, 95% CI 2-sided [-4.50 to 6.70], Standard Error of Mean 2.83

17. Secondary Outcome: Baseline Work Productivity and Activity Impairment (WPAI): Percent Activity Impairment
Description: Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI asks participants about the effect of urinary leakage on their ability to perform their work-related functions and carry out daily activities over the past seven days. Percent activity impairment is derived from the participant's assessment of the degree to which their urinary leakage affected their regular daily activities. A higher percentage indicates greater impairment and less productivity.
Time Frame: Baseline
Population: Full analysis set participants with available WPAI data at Baseline.
Measure: Mean (Standard Deviation); unit: percent activity impairment
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 127 | 147
percent activity impairment | 41.6 (28.38) | 41.4 (27.49)

18. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Activity Impairment
Description: Work productivity was measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). WPAI asks participants about the effect of urinary leakage on their ability to perform their work-related functions and carry out daily activities over the past seven days. Percent activity impairment is derived from the participant's assessment of the degree to which their urinary leakage affected their regular daily activities. A higher percentage indicates greater impairment and less productivity. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set with available WPAI data at both Baseline and each time point; "n" indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: Percent activity impairment
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 124 | 145
Percent activity impairment
  Week 12 (n=115, 129) | -28.2 (1.93) | -30.2 (1.82)
  End of treatment (n=124, 145) | -28.4 (1.95) | -28.8 (1.78)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Comparison at Week 12; Test type: Superiority or Other; p = 0.4067, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 2.0, 95% CI 2-sided [-2.80 to 6.89], Standard Error of Mean 2.46
Statistical Analysis 2: Comparison: Placebo vs Solifenacin Succinate; Comparison of end of treatment analysis; Test type: Superiority or Other; p = 0.8507, ANCOVA; [statistical method as in outcome 6, analysis 1]; Treatment Difference = 0.4, 95% CI 2-sided [-4.21 to 5.10], Standard Error of Mean 2.36

19. Secondary Outcome: Time From Baseline to First Day of Returning to Work
Description: The time from Baseline to first day of returning to work was estimated using the Kaplan-Meier method.
Time Frame: From Baseline to Week 12
Population: Full analysis set participants who were employed prior to the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 127 | 147
days | 5.0 [4.0 to 12.0] | 5.0 [3.0 to 8.0]
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Test type: Superiority or Other; p = 0.2700, Log Rank; Based on a Log-rank test stratified by (pooled) center

ADVERSE EVENTS:
Time Frame: From the first dose of study drug and within 7 days after last dose of study drug (13 weeks).
Arm/Group | Placebo | Solifenacin Succinate
Serious Adverse Events (participants affected / at risk) | 5/310 | 7/313
Other Adverse Events (participants affected / at risk) | 2/310 | 19/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=310) | Solifenacin Succinate (N=313)
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Infected Lymphocele (Infections and infestations) | 0 | 1
Psoas Abscess (Infections and infestations) | 1 | 0
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Lymphocele (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=310) | Solifenacin Succinate (N=313)
Dry mouth (Gastrointestinal disorders) | 2 | 19

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data, or 18 months after data lock, whichever occurs first. Sponsor must receive a site's manuscript at least 30 days prior to publication for review and comment. Sponsor may delay the publication for up to 60 days to seek patent protection.